CLINICAL TRIAL: NCT01438138
Title: Validation of a Classifier for the Prediction of Risk of Relapse Using Single Cell Network Profiling (SCNP) Assays for Childhood AML
Brief Title: Study to Predict Risk of Relapse in Bone Marrow Cell Samples From Younger Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B12; CDR0000711851 (Other: Clinical Trials.gov); COG-AAML11B2 (Other: Children's Oncology Group); NCI-2011-03465 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-17; First posted 2011-09-21 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute basophilic leukemia; childhood acute eosinophilic leukemia; childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Eosinophilic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Archived bone marrow mononuclear cells are analyzed by single cell network proteomic profiling assay, the My Profile™ AML Risk of Relapse Assay. Molecular markers analyzed include Flt3-ITD, NPM1, and MRA. Results are then correlated with each patient's clinical data including patient's age, race/ethnic background, gender, treatment received, and outcomes.
  Interventions: Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: A screening test, such as My Profile Pediatric Assay, may help doctors predict a patient's risk of relapse and plan better treatment for acute myeloid leukemia.

PURPOSE: This clinical trial is studying using the My Profile Pediatric Assay to see how well it works in predicting risk of relapse in bone marrow cell samples from younger patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To validate the accuracy of the My Profile Pediatric Assay to predict risk of relapse in pediatric patients with non-M3 acute myeloid leukemia (AML) who responded to cytarabine-based induction chemotherapy.

Secondary

* To validate the continuous score from the pre-specified classifier as a predictor of relapse after response to induction chemotherapy, while controlling for the simultaneous effects of the following clinical and laboratory variables: age, WBC, ethnicity, cytogenetics, Flt3-ITD, NPM1, MRD, and bone marrow (BM) donor availability.
* To validate the accuracy of the prespecified low versus high relapse indicator variable (I_L/H) as a predictor of relapse after induction therapy.
* To validate the accuracy of the prespecified I_L/H as a predictor of relapse after induction therapy, while controlling for the simultaneous effects of the following clinical and laboratory variables: MRD, age, WBC, ethnicity, cytogenetics, Flt3-ITD, NPM1, and BM donor availability.

OUTLINE: Archived bone marrow mononuclear cells are analyzed by single cell network profile assay, the My Profile™ AML Risk of Relapse Assay. Molecular markers analyzed include Flt3-ITD, NPM1, and MRA. Results are then correlated with each patient's clinical data including patient's age, race/ethnic background, gender, treatment received, and outcomes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with confirmed non-M3 acute myeloid leukemia

  * Treated on COG-AAML03P1 or COG- AAML0531 protocols

    * Samples from COG-AAML0531 can come from either treatment arm, but these samples need to be independent from any patients who donated samples assayed in study COG-AAML11B2
  * Patients with Down syndrome are excluded
* Cryopreserved bone marrow mononuclear cell (BMMC) samples collected at diagnosis, prior to start induction therapy

  * Samples must have been cryopreserved at central lab within 3 days of draw at clinical site
  * Target of 10 X 10^6 cells frozen
* Patients' clinical annotations required after unblinding

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with confirmed non-M3 acute myeloid leukemia treated on COG-AAML03P1 or COG-AAML0531 protocols
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve of continuous score from the pre-specified classifier in predicting relapse after complete response to cytarabine- based induction chemotherapy | Up to 3 years
  A logistic regression model and area under the ROC curve for the model will be tested for significance against a null value of 0.5.

SECONDARY OUTCOMES:
Continuous score from the pre-specified classifier as a predictor of relapse after response to induction chemotherapy | Up to 3 years
  A gate-keeper strategy will be applied to control the experiment-wise type I error rate at 0.05. The null hypothesis will be tested using a likelihood ratio test that will compare the likelihood for a full (LF) and a reduced (LR) logistic regression model of relapse (early relapse vs continuous complete response), where the full model will include the covariates and the continuous score from the pre-specified classifier and the reduced model will include only the covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Norman J. Lacayo, MD, Principal Investigator — Stanford University